CLINICAL TRIAL: NCT03199521
Title: Assessing The Effect of Apixaban on Endogenous Fibrinolysis in Patients With Non-Valvular Atrial Fibrillation
Brief Title: Assessment of The Effect of Apixaban in AF
Status: Completed | Type: Observational
Sponsor: East and North Hertfordshire NHS Trust (Other Government)
Collaborators: University of Hertfordshire (Other)
Responsible Party: Principal Investigator, Prof Diana Gorog, Professor,University of Hertfordshire, East and North Hertfordshire NHS Trust
Other Study IDs: No 1.1 Apr 2017; CV185-622 (Other Grant/Funding Number: BMS/Pfizer European Thrombosis Investigator Initiated Research Program); RD2017-03 (Other: East and North Hertfordshire NHS Trust)
Record Dates: First submitted 2017-06-13; First posted 2017-06-27 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Atrial Fibrillation; Embolism Thrombosis
Keywords: apixaban; endogenous fibrinolysis; warfarin; aspirin; thrombotic status
MeSH Terms: conditions — Atrial Fibrillation; Embolism and Thrombosis | interventions — Thrombelastography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Atrial Fibrillation newly diagnosed, starting apixaban: Patients will undergo the global thrombosis test (GTT), thromboelastography (TEG) and thrombin generation assays before and after stabilisation(4 weeks) of their anticoagulation. This will allow to compare the effect of apixaban on endogenous fibrinolysis before and after treatment.
  Interventions: Other: Thrombin generation assays, Thromboelastography (TEG), and Global Thrombosis Test (GTT)
- Atrial fibrillation on stable warfarin treatment: Patients will undergo the global thrombosis test (GTT), thromboelastography (TEG) and thrombin generation assays on stable anticoagulation treatment. This will allow to compare the effect of apixaban against warfarin on endogenous fibrinolysis on stable treatment.
  Interventions: Other: Thrombin generation assays, Thromboelastography (TEG), and Global Thrombosis Test (GTT)
- Atrial Fibrillation on stable aspirin treatment: Patients will undergo the global thrombosis test (GTT), thromboelastography (TEG) and thrombin generation assays on stable anticoagulation treatment. This will allow to compare the effect of apixaban against aspirin on endogenous fibrinolysis on stable treatment.
  Interventions: Other: Thrombin generation assays, Thromboelastography (TEG), and Global Thrombosis Test (GTT)

INTERVENTIONS:
Other: Thrombin generation assays, Thromboelastography (TEG), and Global Thrombosis Test (GTT) — Global Thrombosis Test (GTT): assesses formation of the blood clot and how easily can this be broken down once formed) Thromboelastography (TEG) :assesses the properties of a blood clot and how easily can be broken down Thrombin generation assays: assesses the formation of a blood clot and the potential of thrombolysis via the introduction of different buffer solutions

SUMMARY:
This study will assess the effect of apixaban on thrombotic status in patients with atrial fibrillation.In addition it will compare apixaban to aspirin and warfarin on their effect on endogenous fibrinolysis.

DETAILED DESCRIPTION:
Patients with an irregular heart rhythm called atrial fibrillation (AF) have an increased risk of forming blood clots inside the heart, that can then fragment and break off, travelling through the circulation to the brain, where it can cause blockage of the small blood vessels resulting in a stroke. Most patients with AF are prescribed blood thinning medications in an attempt to prevent such clot formation. The body has the ability through enzymes circulating in blood, to dissolve a clot once formed, such that even if a clot is formed, it is rapidly dissolved and no lasting damage is sustained. This is known as endogenous fibrinolysis. If this defence system is faulty or suboptimal, there is an increased risk of clot formation, resulting in stroke or heart attack. Currently, there are no available tablets to favourably modify this defence system of endogenous fibrinolysis. The investigators will assess how this defence system functions in patients with AF who are on different blood thinners. Then the investigators will also assess a group of patients before and during treatment with a relatively new blood thinner called apixaban, to assess the effect of this on the stickiness of blood and the ability of the blood to dissolve clots (endogenous fibrinolysis). All the blood thinners will be prescribed for clinical indications, not as part of the research. The research aspect of the study is that we will perform a blood test to assess endogenous fibrinolysis.

Understanding the effect of apixaban on endogenous fibrinolysis raises the possibility that apixaban, rather than other blood thinners, may be of particular use in patients with impaired fibrinolysis who are at particularly high risk of clots due to inefficient endogenous fibrinolysis.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Diagnosis of NVAF (nonvalvular atrial fibrillation)
3. Requiring anticoagulation or antiplatelet therapy for thromboprophylaxis of stroke and systemic embolism
4. No contra-indications to apixaban (except for those patients taking part in baseline cross-sectional study where this inclusion criterion does not apply)
5. Patient does not meet any of the exclusion criteria below

Exclusion Criteria:

1. Patient unwilling or unable to give informed consent
2. Patient already taking antiplatelet or anticoagulant therapy (except for those patients taking part in baseline cross-sectional study, where this exclusion criterion does not apply)
3. Patient who, in the opinion of the investigator, has significant hepatic or renal impairment likely to cause a bleeding diathesis
4. Patient needing systemic high dose steroids or immunosuppression that may impact on platelet function
5. Patient with ongoing active alcohol or substance abuse or demonstrates signs or clinical features of active substance abuse
6. Patient with any major bleeding diathesis or blood dyscrasia at baseline (platelets<70 x 109/l, Hb<80 g/l, INR >1.4 (international normalized ratio), APTT (activated partial thromboplastin time ) > x 2UNL (upper normal limit) , leucocyte count< 3.5x 109/l, neutrophil count<1x 109/l).
7. Patient currently involved in another investigational trial of a medicine or medical device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-valvular atrial fibrillation. Participants will be recruited via inpatient and outpatient clinical areas.
Sampling Method: Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-01-02 (Actual); Study Completion 2019-01-02 (Actual)

PRIMARY OUTCOMES:
Assessing the effect of apixaban on endogenous fibrinolysis in patients wth atrial fibrillation | Change of endogenous fibrinolysis from baseline at 4 weeks
  Measuring endogenous fibrinolysis before and after apixaban

SECONDARY OUTCOMES:
Comparing the effect of apixaban to warfarin and aspirin on endogenous fibrinolysis in patients with atrial fibrillation | 12 months
  Compare the effect on endogenous fibrinolysis as measured by occlusion time and lysis time (seconds) of stable apixaban, warfarin and aspirin treatment in patients with atrial fibrillation with the GTT,TEG,thrombin generation assays

CONTACTS AND LOCATIONS:
Locations (1):
- Hertfordshire Cardiology Centre, East and North Hertfordshire NHS Trust, Stevenage, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes